CLINICAL TRIAL: NCT05805150
Title: Performance Evaluation of Different Daily Disposable Contact Lenses in Habitual Lens Wearers Who Report Frequent Use of Digital Devices
Brief Title: Performance Evaluation of Daily Disposable Contact Lenses in Habitual Lens Wearers Who Use Digital Devices Frequently
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-148
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lens, Then Test Lens (Experimental): Participants will wear control lenses for one week and then crossover to test lenses for one week.
  Interventions: Device: Control Lens (stenfilcon A); Device: Test Lens (senofilcon A)
- Test Lens, Then Control Lens (Experimental): Participants will wear test lenses for one week and then crossover to control lenses for one week.
  Interventions: Device: Control Lens (stenfilcon A); Device: Test Lens (senofilcon A)

INTERVENTIONS:
Device: Control Lens (stenfilcon A) — One week wear
Device: Test Lens (senofilcon A) — One week wear

SUMMARY:
The goal of this study is to compare the performance of two daily disposable silicone hydrogel lenses.

DETAILED DESCRIPTION:
This study is prospective, bilateral eye, double masked, randomized, 1 week cross-over, daily wear design involving in two different daily disposable lens types. Each lens type will be worn for approximately one week.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 35 years of age (inclusively) and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Self-reports having a full eye examination in the previous two years;
* Self-reports spending on most days at least 6 hours cumulative (not necessarily in one single stretch) using digital devices such as a computer, laptop, tablet, e-reader, smartphone;
* Anticipates being able to wear the study lenses for at least 8 hours a day, 7 days a week;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Habitually wears soft contact lenses, for the past 3 months minimum;

  1. No more than 1/3 of participants should be habitual wearer of MyDay or MyDay Energys
  2. No more than 1/3 of participants should be habitual wearer of ACUVUE® OASYS MAX 1-Day or ACUVUE® OASYS 1-Day.
* Has refractive astigmatism no higher than -0.75DC in each eye;
* Can be fit and achieve binocular distance vision of at least 20/30 Snellen (Available lens parameters are sphere -1.00 to -6.00D, 0.25D steps).

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active ocular disease and/or infection that contraindicates contact lens wear;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
* Has known sensitivity to the diagnostic sodium fluorescein used in the study;
* Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
* Has undergone refractive error surgery or intraocular surgery.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Wesley, Principal Investigator — Complete Eye Care of Medina; Michael Cymbor, Principal Investigator — Nittany Eye Associates; Shane Kannarr, Principal Investigator — Kannarr Eye Care; Stephen Montaquila, Principal Investigator — West Bay Eye Associates
Locations (4):
- United States (4):
  - Kannarr Eye Care, Pittsburg, Kansas
  - Complete Eye Care of Medina, Medina, Minnesota
  - Nittany Eye Associates, State College, Pennsylvania
  - West Bay Eye Associates, Warwick, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Lens, Then Test Lens: Participants wore Control Lens for 1 week (Period 1), and then Test Lens for 1 week (Period 2).
- Test Lens, Then Control Lens: Participants wore Test Lens for 1 week (Period 1), and then Control Lens for 1 week (Period 2).
Period: Period 1 (1 Week)
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 34 | 35
Completed | 34 | 35
Not Completed | 0 | 0
Period: Period 2 (1 Week)
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 34 | 35
Completed | 34 | 34
Not Completed | 0 | 1
Not completed — Should not have been enrolled. Participant was nursing (lactating). | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Analysis Population: All participants who completed study. (Total study population n=68)
Arm/Group | Analysis Population
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling on Removal
Description: Ease of lens removal on a 0-100 scale (0= very difficult, 100= very easy)
Time Frame: Collected once on day 6 at the end of wear
Population: Total Analysis Population is 68, only those who completed the study.
Measure: Median (Standard Deviation); unit: Units on a scale
Groups:
- Control Lens: Participants that received Control lens during either the first or second period of the study
- Test Lens: Participants that received Test lens during either the first or second period of the study
Arm/Group | Control Lens | Test Lens
Number analyzed (Participants) | 68 | 68
Units on a scale | 90 (18) | 95 (8)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 2 weeks.
Arm/Group | Control Lens | Test Lens
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 1/69 | 1/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Lens (N=69) | Test Lens (N=69)
Redness and Swelling (Eye disorders) | 0 (0) | 1 (1)
Redness and small bump on lid (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT05805150/Prot_SAP_000.pdf